CLINICAL TRIAL: NCT04019652
Title: A Randomized, Double-Blind, Single-Dose, Placebo- and Positive-Controlled Crossover Study to Evaluate the Effect of Therapeutic and Supratherapeutic Exposure to CS-3150 on QTc Interval Duration in Healthy Male and Female Subjects
Brief Title: The Effect of CS-3150 Exposure on Corrected QT (QTc) Interval Duration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CS3150-A-U106
Record Dates: First submitted 2019-07-09; First posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Hypertension; Mineralocorticoid Receptor Antagonist
Keywords: Hypertension; Mineralocorticoid receptor antagonist
MeSH Terms: conditions — Hypertension | interventions — esaxerenone; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: This is a phase 1, single center, randomized, single-dose, double-blind, double-dummy, placebo- and positive-controlled, 4-period crossover study. Participants will be randomized to one of the following 4 treatment sequences:
  1. CS-3150 (10-mg dose)/CS-3150 (40-mg dose)/moxifloxacin/placebo
  2. CS-3150 (40-mg dose)/placebo/CS-3150 (10-mg dose)/moxifloxacin
  3. Moxifloxacin/CS-3150 (10-mg dose)/placebo/CS-3150 (40-mg dose)
  4. Placebo/moxifloxacin/CS-3150 (40-mg dose)/CS-3150 (10-mg dose)
Who Masked: Participant, Investigator
Masking Description: The Investigator, participants, and all other clinical management and personnel will be blinded to treatment. CS-3150 and moxifloxacin (positive control) treatments will be blinded by matching placebos.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 10 mg CS-3150 (Treatment Sequence 1) (Experimental): Participants will receive the following treatment sequence (1 treatment per Period): a single oral 10-mg dose of CS-3150, a 40-mg dose of CS-3150, a 400-mg dose of moxifloxacin, followed by placebo.
  Interventions: Drug: CS-3150; Drug: Moxifloxacin; Drug: Placebo matching moxifloxacin tablet
- 40 mg CS-3150 (Treatment Sequence 2) (Experimental): Participants will receive the following treatment sequence (1 treatment per Period): a single oral 40-mg dose of CS-3150, placebo, a 10-mg dose of CS-3150, followed by a 400-mg dose of moxifloxacin.
  Interventions: Drug: CS-3150; Drug: Moxifloxacin; Drug: Placebo matching moxifloxacin tablet
- Moxifloxacin (Treatment Sequence 3) (Experimental): Participants will receive the following treatment sequence (1 treatment per Period): a single oral 400-mg dose of moxifloxacin, 10-mg dose of CS-3150, placebo, 40-mg dose of CS-3150.
  Interventions: Drug: CS-3150; Drug: Moxifloxacin; Drug: Placebo matching CS-3150
- Placebo (Treatment Sequence 4) (Experimental): Participants will receive the following treatment sequence (1 treatment per Period): a single oral dose of placebo, 400-mg dose of moxifloxacin, 40-mg dose CS-3150, 10-mg dose of CS-3150.
  Interventions: Drug: CS-3150; Drug: Moxifloxacin; Drug: Placebo matching moxifloxacin tablet; Drug: Placebo matching CS-3150

INTERVENTIONS:
Drug: CS-3150 — Single, oral administration; 10-mg or 40-mg dose
  Other Names: Esaxerenone
Drug: Moxifloxacin — Single, oral administration; 400 mg-tablet
  Other Names: Avelox
Drug: Placebo matching moxifloxacin tablet — Placebo tablets matching moxifloxacin tablets
  Other Names: Placebo
  Arms: 10 mg CS-3150 (Treatment Sequence 1); 40 mg CS-3150 (Treatment Sequence 2); Placebo (Treatment Sequence 4)
Drug: Placebo matching CS-3150 — Placebo tablets matching CS-3150 tablets
  Other Names: Placebo
  Arms: Moxifloxacin (Treatment Sequence 3); Placebo (Treatment Sequence 4)

SUMMARY:
This study will test if a study drug (CS-3150) will affect the heart rate in healthy males and females. Two doses of the study drug will be tested. Heart rate is not expected to be different between the study groups.

DETAILED DESCRIPTION:
This study will assess the effect of therapeutic and supratherapeutic plasma exposures of CS-3150 on the corrected QT (QTc) interval duration after administration of single oral 10-mg and 40-mg doses of CS-3150 in healthy male and female participants. This study will also determine the safety and tolerability of CS-3150 administration, assess the effect on electrocardiogram (ECG) parameters, detect QT interval (QT)/QTc prolongation with a positive control (moxifloxacin), characterize pharmacokinetics (PK) of CS-3150, and assess exposure-response relationship of CS-3150 on QTc.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and/or females 18 years to 45 years of age with a body mass index of 19 kg/m2 to 32 kg/m2 (inclusive)
* Laboratory results (serum chemistry, hematology, and urinalysis [UA]), liver function, and serum K+ levels within normal range
* Written informed consent
* Female participants: Negative pregnancy test and must either be surgically sterile, postmenopausal, or agree to use acceptable nonhormonal contraception.

Exclusion Criteria:

* All prescription or over-the-counter (OTC) medication (systemic and topical) and herbal supplements will not be permitted for 14 days before the first dose and for the duration of the study.
* Oral, injected, or implanted hormonal contraception methods, or hormonal replacement therapy, should not have been received in the 3 months prior to the first dose, and for the duration of the study.
* Female participants: positive pregnancy test or are breast feeding.
* Supine systolic/diastolic blood pressure at screening, after resting for 10 min, higher than 140/90 mmHg or lower than 90/50 mmHg, confirmed after repeated testing at least approximately 1 h apart.
* Supine pulse at screening, after resting for 10 min, outside the range of 40 to 100 beats per minute (bpm).
* QTcF interval duration > 450 ms for male and female obtained as an average from the triplicate screening ECGs after at least 10 min in a fully supine quiet rest.
* Abnormal waveform morphology on any of the screening ECGs that would preclude accurate measurement of the QT interval duration.
* Family history of congenital Long QT syndrome (LQTS), a history of surviving an unexplained drowning episode, a history of any form of syncope or loss of consciousness, or known symptomatic cardiac arrhythmias.
* Known allergy to moxifloxacin.
* An estimated glomerular filtration rate (eGFR) using the Modification of Diet in Renal Disease (MDRD) equation lower than 90 mL/min.
* Previous participation in a CS-3150 study within 6 months prior to the single dose of CS-3150.
* History or current evidence of clinically significant cardiac, hepatic, renal, pulmonary, endocrine, neurologic, infectious, gastrointestinal, hematologic, or oncologic disease as determined by the PI after reviewing screening history, physical examination, laboratory test results, and 12-lead ECG
* Clinically significant illness (at the discretion of principal investigator) within 4 weeks of first dose, are carriers of Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (HCV), or human immunodeficiency virus (HIV) antibody, and any other reason not deemed suitable for the study (at the discretion of the principal investigator).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2015-12-23 (Actual); Study Completion 2015-12-23 (Actual)

PRIMARY OUTCOMES:
Change in corrected QT (QTc) interval from baseline following oral administration of 1 of 4 treatment sequences with CS-3150 | Day -1 of Period 1 through Day 8 of Period 4 (~36 days)
  On the electrocardiogram tracing, the estimated difference in least square means will be reported between each CS-3150 dose level and placebo in QTc change from baseline.

SECONDARY OUTCOMES:
Percentage of participants reporting treatment-emergent adverse events (TEAEs) following oral administration of 1 of 4 treatment sequences with CS-3150 | Day -1 of Period 1 through Day 8 of Period 4 (~36 days)
Change in corrected QT (QTc) interval from baseline following oral administration of 1 of 4 treatment sequences with moxifloxacin | Day -1 of Period 1 through Day 8 of Period 4 (~36 days)
  On the electrocardiogram tracing, the estimated difference in least square means will be reported between moxifloxacin and placebo in QTc change from baseline.
Change in the interval between the P and R waves (PR) from baseline following oral administration of 1 of 4 treatment sequences with CS-3150 | Day -1 of Period 1 through Day 8 of Period 4 (~36 days)
  On the electrocardiogram tracing, the interval between the P and R waves (PR) at baseline and change from baseline will be summarized by treatment.
Change in QRS wave complex (QRS) from baseline following oral administration of 1 of 4 treatment sequences with CS-3150 | Day -1 of Period 1 through Day 8 of Period 4 (~36 days)
  On the electrocardiogram tracing, QRS wave complex (QRS) at baseline and change from baseline will be summarized by treatment.
Change in QT interval (QT) from baseline following oral administration of 1 of 4 treatment sequences with CS-3150 | Day -1 of Period 1 through Day 8 of Period 4 (~36 days)
  On the electrocardiogram tracing, QT interval (QT) at baseline and change from baseline will be summarized by treatment.
Change in QTc corrected by Bazett's formula (QTcB) from baseline following oral administration of 1 of 4 treatment sequences with CS-3150 | Day -1 of Period 1 through Day 8 of Period 4 (~36 days)
  On the electrocardiogram tracing, QTc corrected by Bazett's formula (QTcB) at baseline and change from baseline will be summarized by treatment.
Change in QTc corrected by Fridericia's formula (QTcF) from baseline following oral administration of 1 of 4 treatment sequences with CS-3150 | Day -1 of Period 1 through Day 8 of Period 4 (~36 days)
  On the electrocardiogram tracing, QTc corrected by Fridericia's formula ([QTcF]) at baseline and change from baseline will be summarized by treatment.
Change in heart rate (HR) from baseline following oral administration of 1 of 4 treatment sequences with CS-3150 | Day -1 of Period 1 through Day 8 of Period 4 (~36 days)
  Based on the electrocardiogram tracing, heart rate (HR) at baseline and change from baseline will be summarized by treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Mendell J, Kobayashi F, Shimizu T. Randomized, Double-Blind, Single-Dose, Placebo-Controlled Crossover Study to Evaluate the Effects of Esaxerenone on QTc Interval in Healthy Subjects. Clin Pharmacol Drug Dev. 2020 Aug;9(6):709-718. doi: 10.1002/cpdd.794. Epub 2020 Apr 7. PMID 32255542